CLINICAL TRIAL: NCT01020695
Title: QEEG and LORETA Analysis in PTSD Patients
Brief Title: Quantitative Electroencephalography (QEEG) and Low-resolution Electromagnetic Tomography (LORETA) Analysis in Post Traumatic Stress Disorder (PTSD) Patients
Status: Completed | Type: Observational
Sponsor: Beersheva Mental Health Center (Other Government)
Responsible Party: Principal Investigator, Doron Todder, Dr., Beersheva Mental Health Center
Other Study IDs: BHC-4917
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD; EEG; QEEG; LORETA
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- PTSD veterans: 18 PTSD veterans
- controls: 20 controls

SUMMARY:
In this study the Quantitative Electroencephalography and low resolution topographic analysis of chronic Post-traumatic stress disorder and normal subjects will be compared.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is defined as a constellation of symptoms in response to a stressor, including re-experiencing a traumatic event, numbed responsiveness and symptoms of an increased level of arousal (APA 2000) . In recent years there were many attempts to connect the brain structure and function to symptoms in PTSD patients (Francati, Vermetten et al. 2007; Liberzon and Sripada 2008). One of the important technologies in this regard is the Electroencephalography (EEG) measurement.

The EEG is the reflection of the inner brain electrical changing dipole as it is measured on the scalp. It is measured by electrode that placed on the head according to the international distribution of electrodes called 10-20. The EEG recording that is the product of the measurement can be analyzed at least in three different levels: visual inspection of the raw EEG, quantities analysis of the EEG (QEEG) and based on the QEEG, calculating the electrical distribution of dipoles inside the brain that creates the EEG signal (Niedermeyer and Lopes da Silva 2005). Theoretically two EEG measurements could have the same visual EEG and/or QEEG patterns but the inner brain electrical dipole distribution could be very different. The mathematical solution to the calculation of the dipole distribution inside the brain, using the scalp EEG is based on "the inverse problem" concepts. One of the more common and precise method to solve the inverse problem regarding the EEG is called LORETA (low resolution topographic analysis) (Pascual-Marqui, Michel et al. 1994; Pascual-Marqui, Esslen et al. 2002). There are many brain image technologies aiming on mapping the connection between brain function and psychopathology. Each method caries with it both advantage and drawbacks. The use of the Electroencephalographic mapping technique is no different and it's main advantage - the temporal resolution is with opposition to the relatively lower spatial resolution. Modern signal processing tools and software like the LORETA start challenging this equation and in the last years some articles were published proving the possibilities of using EEG measurement to localized brain function with high spatial-resolution (Stern, Neufeld et al. 2009) .

The study will focus on the rest QEEG and rest LORETA analysis in PTSD patients.

Previous QEEG research found conflicting results regarding the spectral distribution of the EEG waves across the scalp.

Begic et al (Begic, Hotujac et al. 2001) compared 18 PTSD veterans to 20 controls. They found that PTSD patients had increased theta activity over central regions, and they had increased beta activity over frontal, central and occipital regions. No significant differences were noted between the PTSD and control group in both the delta and alpha activity. In this study all the patients were medication free for 2 weeks.

In another study the same group compared veterans with PTSD to veterans without PTSD. In this study the PTSD patients had decreased alpha power and increased beta power. No difference was noted on the theta band in this study (Jokic-Begic and Begic 2003).

In a recent study another group studied the hemispheric asymmetries among motor vehicle survivors with PTSD, with subsyndromal PTSD, survivors without PTSD and nonexposed healthy controls during rest (baseline) and in response to neutral, positive, negative, and trauma-related pictures. They focus on the alpha band. They found no group differences in EEG alpha activity during the baseline condition. In there study all the patients were without medication for 1 month (Rabe, Beauducel et al. 2006). Shankman et al compared the resting EEG of PTSD patients to "super- controls" in order to maximized the difference between this two groups. They found no statistical significant difference in any of the spectral band (Shankman, Silverstein et al. 2008).

The aim of this study is to calculate the QEEG difference and to do LORETA analysis in PTSD patients compared to controls.

In order to avoid statistical multiple compressing problems this study will focus on the theta band. There are at least two reasons for this: the first is that due to ethical issue we don't ask our patients to stop there psychotropic treatments therefore all of them are using SSRI antidepressants which could cause some alpha rhythms changes (Niedermeyer and Lopes da Silva 2005). Another reason is that the origin of the theta bend is supposed to be the in limbic system (Niedermeyer and Lopes da Silva 2005) that is long ago connected to PTSD symptoms (Francati, Vermetten et al. 2007).

ELIGIBILITY:
Inclusion Criteria:

* 10 veterans suffering for PTSD according to the DSM-IV-TR for at least 2 years.
* The 10 age matching controls will be recruited from the Beer Sheva mental stuff.

Exclusion Criteria:

* Without any neurological or head trauma.
* Without alcohol or substance abuse.
* No evidence of psychotic episode in there history.
* Stable doses of different specific serotonin reuptake inhibitors (SSRI) antidepressant for at least two months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Veterans with chronic PTSD of at least 2 years.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Beer Sheva Mental Health Center, Beersheba, Israel